CLINICAL TRIAL: NCT05472103
Title: Strategies for Musculoskeletal Symptoms Relieving and Ergonomy in Operating Room: a Prospective Clinical Trial. (MuSEO Study)
Brief Title: Strategies for Musculoskeletal Symptoms Relieving and Ergonomy in Operating Room
Acronym: MuSEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof. Antonino Agrusa, Full Professor of Surgery, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MuSEO study
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Musculoskeletal Pain; Surgery
Keywords: Musculoskeletal Pain; ergonomics; surgery
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): administration of Surgical ergonomics workshop
  Interventions: Behavioral: ergonomics surgical workshop
- control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: ergonomics surgical workshop — ergonomics surgical workshop
  Arms: treatment

SUMMARY:
It is well known that surgery requires not only a mental diligence, but also a real physical stress due to the need to assume particular postures for many hours or to repeat specific maneuvers several times. To this peculiar condition of surgical specialities over the years has been added the development of a series of instruments and technologies ranging from the use of loopes, to laparoscopic and robotic surgery. From the studies reported in the literature, between 74% and 87% of surgeons report symptoms related to their work with consequent effects on the quality of life (sleep loss, inability to carry out their recreational activities, etc.). Similarly, a lack of knowledge of the principles of ergonomics to be applied during the performance of one's surgical activity emerged, which could improve musculoskeletal symptoms with a positive effect on the quality of life of surgeons and consequently hoping for an improvement in professional performance.

ELIGIBILITY:
Inclusion Criteria:

* young surgeons

Exclusion Criteria:

* no consent to partecipate

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-10 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
rate of musculoskeletal symptoms | one month

SECONDARY OUTCOMES:
quality of life | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Giuseppe Di Buono, Palermo, PA, Italy

IPD SHARING:
Plan to Share IPD: No